CLINICAL TRIAL: NCT07065851
Title: Comparison of the Effects of Extracorporeal Shock Wave Therapy and Exercise on Pain, Flexibility, and Balance in Individuals With Hamstring Tightness
Brief Title: Comparison of Shockwave Therapy and Exercise on Pain, Flexibility, and Balance in Hamstring Tightness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Mitra Valaei Bakhshayesh, Principal Investigator,MSc Student in Physiotherapy and Rehabilitation, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bah-YLTez25
Record Dates: First submitted 2025-06-05; First posted 2025-07-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain; Hamstring Tightness
Keywords: Low back pain; Hamstring tightness; Flexibility; Balance; Exercise; Shock wave therapy; Extracorporeal Shock Wave Therapy (ESWT)
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Extracorporeal Shockwave Therapy; Resistance Training

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment model with two intervention arms. Thirty participants with low back pain related to hamstring tightness are randomly assigned to two groups (n=15 each): extracorporeal shock wave therapy (ESWT) or exercise therapy. Interventions are delivered 1-2 times per week for four weeks. The ESWT group receives standardized shock wave therapy targeting the hamstring muscles. The exercise group follows a structured program including hamstring stretching, lumbar stabilization, and core exercises. Participants remain in their assigned groups throughout the study with no crossover. Outcome measures-pain intensity (Visual Analog Scale), hamstring flexibility (Popliteal Angle and Fingertip-to-Floor tests), and dynamic balance (Y-Balance Test)-are assessed at baseline, post-intervention (week 4), and follow-up (week 8). Single blinding is applied for the outcome assessor to minimize bias in measurements.
Who Masked: Outcomes Assessor
Masking Description: This study employs single blinding, where outcomes assessors are masked to participants' group assignments. Thirty participants are randomized into two groups (extracorporeal shock wave therapy or exercise therapy), with interventions administered by unblinded study personnel. To minimize bias, assessors measuring outcomes, including pain intensity (Visual Analog Scale), hamstring flexibility (Popliteal Angle and Fingertip-to-Floor tests), and dynamic balance (Y-Balance Test), are unaware of the intervention each participant receives. Participants and intervention providers are not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT Group (Experimental): Participants in this group will receive ESWT two times per week for 4 weeks. The treatment will target hamstring muscles and related structures using a standardized ESWT protocol (fixed frequency, intensity, and session duration). In addition to ESWT, participants will perform core strengthening exercises during each session.
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)
- Exercise Group (Active Comparator): Participants in this group will perform a structured exercise program three times per week for 4 weeks. Each session will last 30-45 minutes and will include hamstring stretching, lumbar stabilization, and core strengthening exercises.
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (ESWT) — Non-invasive therapy delivering high-energy shock waves to stimulate healing in musculoskeletal tissues, targeting the hamstring muscles and related structures, administered 2 times per week for 4 weeks, alongside core exercises.
  Arms: ESWT Group
Behavioral: Exercise Program — Structured exercises focusing on hamstring flexibility, lumbar stabilization, and core exercises, administered 3 times per week for 3 weeks, with sessions lasting 30-45 minutes.
  Arms: Exercise Group

SUMMARY:
This randomized controlled trial aims to compare the short- and long-term effects of extracorporeal shock wave therapy (ESWT) and exercise therapy on pain, flexibility, and balance in individuals with low back pain associated with hamstring tightness. Thirty participants will be randomized into two groups (ESWT or exercise) and receive interventions twice weekly for four weeks. Outcomes include pain (a (VAS), flexibility (Popliteal Angle and Fingertip-to-Floor tests), and balance (Y-Balance Test), assessed at baseline, post-intervention, and at a four-week follow-up.

DETAILED DESCRIPTION:
This study evaluates the efficacy of ESWT versus exercise therapy in managing low back pain due to hamstring tightness. Participants with diagnosed hamstring tightness and low back pain will be randomly assigned to receive either ESWT or an exercise program, each administered twice weekly for four weeks. The ESWT group will receive standardized shock wave therapy targeting the hamstring muscles and related structures, alongside core exercises. The exercise group will perform a structured program including hamstring stretching and lumbar stabilization exercises, also with core exercises. Assessments will occur at baseline, immediately post-intervention, and four weeks post-treatment. Pain will be measured using the Visual Analog Scale (VAS), flexibility via Popliteal Angle (PA) and Fingertip-to-Floor (FTF) tests, and balance using the Y-Balance Test (YBT). Data will be analyzed using Statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS), 26.0, with a significance level of p<0.05. The study hypothesizes that ESWT may provide faster pain relief and balance improvements, while exercise may offer more sustained flexibility gains.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed with low back pain due to hamstring tightness.

  * Aged 18-65 years.
  * Male or female.
  * Medically cleared for ESWT or exercise therapy.
  * Experienced low back pain in the past 6 months without serious spinal pathology (e.g., herniated disc, fracture).

Exclusion Criteria:

* • Other musculoskeletal conditions causing low back pain (e.g., disc herniation, spinal stenosis).

  * Outside the specified age range.
  * Serious health conditions that may affect study outcomes.
  * Pregnant or breastfeeding women.
  * Surgical intervention in the back or hamstring region within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, Week 4 (Post-treatment), Week 8 (Follow-up)
  Measured using the Visual Analog Scale (VAS), a 0-10 scale where 0 indicates no pain and 10 indicates the worst imaginable pain.
Hamstring Flexibility (Popliteal Angle) | Baseline, Week 4 (Post-treatment), Week 8 (Follow-up)
  Measured using the Popliteal Angle Test with a goniometer in degrees to assess hamstring muscle flexibility.
Hamstring Flexibility (Fingertip-to-Floor Distance) | Baseline, Week 4 (Post-treatment), Week 8 (Follow-up)
  Measured in centimeters as the vertical distance between the fingertip and the floor during a forward bend with knees extended.
Dynamic Balance (Y-Balance Test) | Baseline, Week 4 (Post-treatment), Week 8 (Follow-up)
  Measured in centimeters using the Y-Balance Test in anterior, posteromedial, and posterolateral directions.

CONTACTS AND LOCATIONS:
Overall Officials: Hasankerem Alptekin, Prof.Dr, Study Director — Bahçeşehir University
Locations (1):
- Bahcesehir University, Istanbul, Healthy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mani-Babu S, Morrissey D, Waugh C, Screen H, Barton C. The effectiveness of extracorporeal shock wave therapy in lower limb tendinopathy: a systematic review. Am J Sports Med. 2015 Mar;43(3):752-61. doi: 10.1177/0363546514531911. Epub 2014 May 9. PMID 24817008
- [Result] Schmitz C, Csaszar NB, Rompe JD, Chaves H, Furia JP. Treatment of chronic plantar fasciopathy with extracorporeal shock waves (review). J Orthop Surg Res. 2013 Sep 3;8:31. doi: 10.1186/1749-799X-8-31. PMID 24004715
- [Result] Rompe JD, Hope C, Kullmer K, Heine J, Burger R. Analgesic effect of extracorporeal shock-wave therapy on chronic tennis elbow. J Bone Joint Surg Br. 1996 Mar;78(2):233-7. PMID 8666632

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT07065851/Prot_SAP_ICF_000.pdf